CLINICAL TRIAL: NCT00939107
Title: The Effect of the McKenzie Method as Compared With That of Manipulation When Applied Adjunctive to Information and Advice for Patients With Clinical Signs of Disc-related Chronic Low Back Pain: Randomized Controlled Trial.
Brief Title: The McKenzie Method Versus Manipulation for Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Back and Rehabilitation Center, Copenhagen (Other Government)
Collaborators: The Danish Rheumatism Association (Other); The Danish Physiotherapy Organization. (Unknown); Foundation for Chiropractic Research and Post Graduate Education (Other); The Danish Institute for Mechanical Diagnosis and Therapy. (Unknown)
Responsible Party: Tom Petersen, research physical therapist, Back and Rehabilitation Center, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KF-01-057/03
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Low Back Pain
Keywords: low back pain; Intervertebral disc; McKenzie; Physical Therapy; Spinal manipulation; Chiropractics; Patient education; Exercise therapy; Random allocation
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- McKenzie exercises (Experimental): McKenzie exercises according to the principles of Mechanical Diagnosis and Therapy
  Interventions: Procedure: McKenzie exercises
- Spinal manipulation (Active Comparator): Spinal manipulation in combination with information of clinical findings and advice about back care
  Interventions: Procedure: spinal manipulation

INTERVENTIONS:
Procedure: spinal manipulation — Spinal manipulation to the lumbopelvic spine in combination with information about examination findings and advice about back care
  Arms: Spinal manipulation
Procedure: McKenzie exercises — McKenzie exercises according to the principles of Mechanical Diagnosis and Therapy
  Arms: McKenzie exercises

SUMMARY:
Introduction:

The McKenzie method as well as spinal manipulation is commonly used for the treatment of low back pain throughout the western world. Recently, the need for studies testing the effect of treatment strategies to specific diagnostic subgroups of patients has been emphasized. The present study aims to compare the effectiveness of the McKenzie method and chiropractic manipulation, information, and advice for patients with clinical signs of persistent symptoms originating from a diskus in the low back.

Methods:

After clinical screening 350 patients with or without leg pain who presented with centralization of symptoms or signs of disc herniation were randomized to the McKenzie group or the manipulation group. The outcome measures, Roland Morris Disability Questionnaire, 11 point numerical pain scale, 6 point global perceived change scale, and quality of life (Short Form-36) were assessed at baseline, at end of treatment, and at 2 and 12 months follow-up.

DETAILED DESCRIPTION:
In 1998, Cherkin et al. published a study showing no difference between outcomes following the McKenzie method, chiropractic manipulation, or the provision of an educational booklet for the treatment of patients with acute non-specific low back pain. Recently, the need for studies testing the effect of treatment strategies to specific diagnostic subgroups of patients has been emphasized. The present study aims to compare the effectiveness of the McKenzie method and chiropractic manipulation, information, and advice for patients with clinical signs of disc-related symptoms for duration of more than 6 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* suffering from low back pain (LBP) with or without leg pain for a period of more than 6 weeks
* able to speak and understand the Danish language
* with a presentation of clinical signs of disc-related symptoms.

Exclusion Criteria:

* positive non-organic signs
* serious pathology suspected based on physical examination and/or magnetic resonance imaging
* application for disability pension or pending litigation
* pregnancy
* comorbidity
* recent back surgery
* problems with communication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2003-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Petersen, PT,PhD, Principal Investigator — Back and Rehabilitation Center Copenhagen, Copenhagen, Denmark
Locations (1):
- Back and Rehabilitation Center Copengagen, Copenhagen, Copenhagen OE, Denmark

REFERENCES:
- [Derived] Petersen T, Christensen R, Juhl C. Predicting a clinically important outcome in patients with low back pain following McKenzie therapy or spinal manipulation: a stratified analysis in a randomized controlled trial. BMC Musculoskelet Disord. 2015 Apr 1;16:74. doi: 10.1186/s12891-015-0526-1. PMID 25887046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients from September 2003 through May 2007 among those referred for treatment at a primary care specialist centre in Copenhagen, Denmark.
Pre-assignment Details: 1969 Patients were screened for eligibility. 1619 Were excluded (580 Were unable to speak and understand Danish, 252 Had comorbidity, 224 Had no peripheralization or centralization, 101 Had previous surgery, 87 Could not be examined, 165 other reasons, 210 Declined to participate)
Period: Overall Study
Arm/Group | McKenzie Exercises | Spinal Manipulation
Started | 175 | 175
12 Months Follow-up | 161 | 163
Completed | 161 | 163
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | McKenzie Exercises | Spinal Manipulation | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 175 | 175 | 350
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (10.4) | 37 (9.4) | 37 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 92 | 195
  Male | 72 | 83 | 155
Region of Enrollment [Number; unit: participants]
  Denmark | 175 | 175 | 350
Number sick-listed [Number; unit: participants]
  Number of patients on sick leave due to LBP | 65 | 47 | 112
  Number of patients not on sick leave due to LBP | 110 | 128 | 238
Duration of pain [Mean (Standard Deviation); unit: Weeks] | 97 (230) | 94 (181) | 95 (210)

OUTCOME MEASURES:

1. Primary Outcome: Disability
Description: Problems performing daily activities measured on the 23-item modified Roland Morris Disability Questionnaire (worst: 23 points, best:0 points).
Time Frame: two months after treatment
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | McKenzie Exercises | Spinal Manipulation
Number analyzed (Participants) | 175 | 175
Units on a scale | 6.7 [5.8 to 7.6] | 5.2 [4.3 to 6.1]
Statistical Analysis 1: Comparison: McKenzie Exercises vs Spinal Manipulation; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Net) = 1.5, 95% CI [0.2 to 2.8]

2. Secondary Outcome: Pain
Description: The back and leg pain questionnaire included three separate 11 point box scales comprising the following items: Low Back Pain (LBP) at the moment, the worst LBP within the past two weeks, and the average level of LBP within the last two weeks. These summed to a total score ranging from 0 points (no back or leg pain at all) to 60 points (worst possible back and leg pain on all items).
Time Frame: twelve months posttreatment
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | McKenzie Exercises | Spinal Manipulation
Number analyzed (Participants) | 175 | 175
Units on a scale | 15.0 [12.9 to 17.1] | 12.2 [10.1 to 14.3]

3. Secondary Outcome: Number of Patients on Sick Leave
Description: Measured by self-report of beeing on sick leave at the moment because of LBP
Time Frame: twelve months posttreatment
Population: Number of patients on sick leave due to LBP pre-treatment.
Measure: Number; unit: Participants
Arm/Group | McKenzie Exercises | Spinal Manipulation
Number analyzed (Participants) | 66 | 47
Participants | 14 | 6

4. Secondary Outcome: Quality of Life
Description: Quality of life, general health, measured on the Short Form 36 questionnaire (worst:100, best:0)
Time Frame: twelve months posttreatment
Reporting Status: Not Posted, anticipated posting 2010-08
Measure: Mean (95% Confidence Interval); unit: Units on a scale

5. Secondary Outcome: Cost Effectiveness
Time Frame: twelve months posttreatment
Reporting Status: Not Posted, anticipated posting 2010-08

6. Primary Outcome: Number of Patients With Treatment Success
Description: Treatment success was defined as a reduction of at least 5 points or an absolute score below 5 points on the 23-item modified Roland Morris Disability Questionnaire (best value: 0 points, worst value 23 points)
Time Frame: Two months posttreatment
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | McKenzie Exercises | Spinal Manipulation
Number analyzed (Participants) | 175 | 175
participants | 120 | 95

ADVERSE EVENTS:
Time Frame: During the intervention which had a duration of maximum 3 months
Description: Adverse events were collected by registration of patients referred to hospital by a rheumatologist due to signs and symptoms of spinal pathology. It is the judgment of the investigators that they were not likely to be provoked by the treatment itself, since treatment currently was guided by the patient's response of symptoms during treatment.
Arm/Group | McKenzie Exercises | Spinal Manipulation
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 5/175 | 9/175
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | McKenzie Exercises (N=175) | Spinal Manipulation (N=175)
herniated disc (Musculoskeletal and connective tissue disorders) | 5 | 9 — Patients referred to hospital due to signs and symptoms of herniated disc by decision of a rheumatologist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes